CLINICAL TRIAL: NCT02639741
Title: Comparison Of The Effects Of Preoperative Melatonin Or Vitamin C Administration On Postoperative Analgesia
Brief Title: Preoperative Melatonin or Vitamin C Administration on Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hakki Unlugenc, Clinical Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZLTNS99
Record Dates: First submitted 2015-11-11; First posted 2015-12-24 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain
Keywords: Melatonin; Vitamin C; Morphine consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Melatonin; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral Melatonin Tablet (Active Comparator): Melatonin, Vitamin C and placebo tablet Preoperative single oral dose of melatonin (6 mg) or placebo tablet will be given one hour before the start of anesthesia.
  Interventions: Drug: Melatonin; Drug: Vitamin C; Other: Placebo
- Oral Vitamin C Tablet (Active Comparator): Melatonin, Vitamin C and placebo tablet Preoperative single oral dose of vitamin C (2 gr) or placebo tablet will be given one hour before the start of anesthesia.
  Interventions: Drug: Melatonin; Drug: Vitamin C; Other: Placebo
- Oral Placebo Tablet (Placebo Comparator): Preoperative single oral dose of placebo tablet will be given one hour before the start of anesthesia.
  Interventions: Drug: Melatonin; Drug: Vitamin C; Other: Placebo

INTERVENTIONS:
Drug: Melatonin — Preoperative melatonin tablet will be given and postoperative pain scores will be evaluated
  Other Names: Melatonina 3 mg tb,
Drug: Vitamin C — Preoperative vitamin C tablet will be given and postoperative pain scores will be evaluated
  Other Names: Vitamin C 1000 mg tb
Other: Placebo — Preoperative placebo tablet will be given and postoperative pain scores will be evaluated
  Other Names: Placebo tb

SUMMARY:
The investigators designed a randomized double-blind placebo-controlled trial to evaluate the effect of preoperative single dose of oral melatonin and vitamin C administration on postoperative analgesia in patients undergoing elective major abdominal surgery.

DETAILED DESCRIPTION:
The investigators designed a randomized double-blind placebo-controlled trial to evaluate the effect of preoperative single dose of oral melatonin and vitamin C administration on postoperative analgesia in patients undergoing elective major abdominal surgery. One hundred-sixty five ASA I-II adult patients between 18-65 years of age, undergoing elective major abdominal surgery with general anesthesia will be included in this double blinded, randomised, controlled study. Patients will randomly divided into equal (n=55) three groups. Preoperatively, one hour before surgery, patients will receive melatonin (6 mg) in group M, vitamin C (2 gr) in group C or placebo tablet in group P orally. A standard anesthetic protocol will be administered to all patients. At the end of surgery, postoperative pain control will be provided via a patient controlled analgesia (PCA) device including morphine in all groups. Hemodynamic parameters, pain, sedation, patient satisfaction, total morphine consumption, supplement analgesic requirement, incidence of nausea and vomiting and other side effects will be recorded at 5, 10, 30 min and 1, 2, 4, 6, 8, 12, 24 hr after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective major abdominal surgery with general anesthesia

Exclusion Criteria:

A history of psychiatric disorders, chronic pain syndromes, obstructive sleep apnea, severe asthma, chronic obstructive pulmonary disease, congestive heart failure, hepatic or renal failure, patients with pregnancy or in lactation period or a history of allergic reaction to any drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-11; Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
morphine consumption at 24 hours after surgery.) | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Hakkı Ünlügenç, Prof Dr., Study Director — Cukurova University
Locations (1):
- Hakkı Ünlügenç, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No